CLINICAL TRIAL: NCT01603316
Title: Food: A Three-Arm Randomized Controlled Study Examining Food Insecurity Interventions
Brief Title: Food: A Three-Arm Study Examining Food Insecurity Interventions
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Queens Cancer Center of Queens Hospital (Other); The Brooklyn Hospital Center (Other); Lincoln Medical and Mental Health Center (Other); Jacobi Medical Center (Other); St. Barnabas Medical Center (Other); Montefiore Health System (Unknown); Columbia University (Other); Roswell Park Cancer Institute (Other); NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 12-099
Record Dates: First submitted 2012-05-16; First posted 2012-05-22 (Estimated); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Cancer Patients
Keywords: Food pantry; Food voucher; Grocery delivery; 12-099
MeSH Terms: interventions — Surveys and Questionnaires; Focus Groups

ARMS (3):
- Food Voucher Program (Voucher) (Active Comparator): Food Voucher arm, each participant will receive a debit card specifically created for this program. Each month for the duration of study participation (6 months), the debit card will be credited with $128 & given to the patient in person or via mail. Patients will be instructed to use these cards only for food purchases. If patients are not able to use the debit card at their local grocery stores, patients will be provided with a money order of the same dollar value instead of the debit card. They will be counseled on using their vouchers only for healthful foods, in a way that stretches their food dollars. Purchases will be tracked by having patients bring their receipts in for review each month when they come in to pick-up their next monthly vouche, or by providing electronic copies of receipts. Patients will be provided with a receipt holder to assist in storing receipts for review. For voucher cards sent via mail, patients will receive a mailing letter accompanying each card.
  Interventions: Behavioral: surveys; Behavioral: Focus groups
- Home Grocery Delivery (Delivery) (Experimental): In the Home Grocery Delivery arm, each participant will receive home grocery delivery from PeaPod grocery delivery service or from FreshDirect (depending on the participant"s zip code), worth $128 per month, for the duration of study participation (6 months). Patients in the Delivery arm will review a list of food categories and a subset of items in each category with a COA.
  Interventions: Behavioral: surveys; Behavioral: Focus groups
- Medically-Tailored Hospital-Based Food Pantry (Pantry) (Experimental): Patients in this arm will have access to the pantry for the duration of their study participation (6 months). Those accessing the medically-tailored food pantry will pick-up a pantry bag weekly or bi-weekly (per patient preference) at the hospital, either during one of their medical appointments or at another preferred time. Each patient's food prefereces will be assessed once during baseline and they will be given food bags, tailored when possible and when available to these preferences and to their medical needs and cultural preferences.
  Interventions: Behavioral: surveys; Behavioral: Focus groups

INTERVENTIONS:
Behavioral: surveys — Each survey will take about 45 minutes.Surveys will include questions on medical treatment, health insurance, work-related information, overall health and well being, eating habits, and satisfaction/use of the food program provided. 3 and 6-month follow-up. All participants will be asked to complete the study contact form. Need Assessment surveys will be administered via telephone or in person. The content of the needs assessment questionnaire has been informed by themes generated through IHCD's ongoing research and community outreach and service activities with the cancer patient population at our participating institutions. The survey will ask participants about the impact on their cancer care and their socioeconomic needs of the COVID-19 crisis.
Behavioral: Focus groups — Prior to conducting the updated RCT design with the expanded cohort, we will conduct 4-6 focus groups (to saturation) with underserved breast cancer patients to optimally tailor the written materials, via mail, MSK Secure email, or in person and nutrition education sessions.

SUMMARY:
The investigators have found that many patients getting treatment for cancer have trouble getting enough to eat, or do not always have enough money for food. When a patient has these problems it can lead to difficulties with completing cancer treatment. Across New York City, there are many hospitals that offer their patients food pantry services on location. The investigators would like to compare how food pantries within the hospital and two other food assistance options: monthly food vouchers and weekly grocery deliveries maybe possible solutions to this problem. The patient will be randomly assigned to one of the three different food program groups, which means everyone has an equal chance in being in any group, like a flip of a coin. The investigators hope to learn how to best help patients with trouble getting food and to see if this will help with completing cancer treatment.

The original RCT composed of study arms: 1) hospital -based food pantry (control), 2) food voucher program plus access to the food pantry, and 3) grocery delivery program plus access to the food pantry will remain open to accrual at Ralph Lauren Cancer Center. The other three sites of the original RCT, Lincoln Hospital, Queens Cancer Center and Brooklyn Hospital, have reached target accrual. Our modified RCT, to be carried out among an expanded cohort of cancer patients is composed of study arms : 1) Food Voucher Program (Voucher); 2) Home Grocery Delivery Program (Delivery); and 3) Medically-tailored, Hospital-based Food Pantry (Pantry).

For this RCT, we will enroll patients across Bronx hospitals- Jacobi Medical Center, St. Barnabas Hospital, and Montefiore Medical Center. For the new study arms, we will enroll patients across Lincoln Medical and Mental Health Center, Jacobi Medical Center, St. Barnabas Medical Center, Montefiore Health System, New York Cancer & Blood Before Specialists, and Bellevue Hospital. Before conducting the RCT across Lincoln Medical and Mental Health Center and the new sites in the Bronx, we will refine written educational materials to be used in the intervention through focus groups.

ELIGIBILITY:
Inclusion Criteria:

Focus Groups Inclusion Criteria:

* Breast cancer patient, Stage 1,2, or 3
* Currently undergoing treatment with chemotherapy and/or radiation
* Food insecure: score in the range of "very low" or "low" food security status on the USDA Household Food Security Module (score of 3 or higher)
* Language spoken: English or Spanish
* Age 18 or over

Intervention Inclusion Criteria:

* Enrolled in ICCAN (for the original arms only: pantry only, pantry + delivery, pantry + voucher)
* Within one month (+/- 1 month) of starting chemotherapy or within two weeks (+/- 2 weeks) of starting radiation therapy) (may be prior to or after starting treatment)
* Score in the range of 'very low' or 'low' food security status on the USDA Household Food Security Module (score of 3 or higher)
* Living independently (no patient in an assisted living facility)
* Age 18 or over
* Able to provide informed consent and respond to questionnaires in either English, Spanish or Mandarin (Mandarin for the original arms only: pantry only, pantry + delivery, pantry + voucher)
* Breast or gynecologic cancer diagnosis, Stage 1, 2, or 3 (for the updated arms only: 1) Food Voucher Program (Voucher); 2) Home Grocery Delivery Program (Delivery); and 3) Medically-tailored, Hospital-based Food Pantry (Pantry)

Clinician is eligible if he/she:

* Has an MD or DO degree
* Is the treating physician providing care to a patient enrolled to the study

Secondary Aim 6 Needs Assessment eligibility criteria:

* Current or past breast cancer diagnosis
* Living independently (no patient in an assisted living facility)
* Age 18 or over
* Able to provide informed consent and respond to questionnaires in either English, or Spanish

Exclusion Criteria:

Focus Groups Exclusion Criteria:

* Has a household member who has already participated (or agreed to participate)

Intervention Exclusion Criteria:

* Significant psychiatric disturbance verified by medical record sufficient to preclude completion of the assessment measures, interview or informed consent (i.e. acute psychiatric symptoms which require individual treatment)
* Presence of cognitive impairment disorder (i.e. delirium or dementia) sufficient to preclude meaningful informed consent and/or data collection
* Can not speak English, Spanish or Mandarin (Mandarin for the original arms only: pantry only, pantry + delivery, pantry + voucher)
* Has physical limitations that would prevent participation (e.g. blindness)
* Patient's household is currently receiving or applying for SNAP benefits (formerly known as Food Stamps) (for the original arms only: pantry only, pantry + delivery,pantry + voucher)

Secondary Aim 6 Needs Assessment Exclusion criteria:

* Significant psychiatric disturbance verified by medical record enough to preclude completion of the assessment measures, interview or informed consent (i.e. acute psychiatric symptoms which require individual treatment)
* Presence of cognitive impairment disorder (i.e. delirium or dementia) enough to preclude meaningful informed consent and/or data collection
* Cannot speak English or Spanish
* Has physical limitations that would prevent participation (e.g. blindness)
* Patient or family member has participated in other MSK IHCD trials related to social determinants of health

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 606 (Actual)
Dates: Start 2012-05-08 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
treatment completion | 2 years
  Completion of prescribed treatment, increase from 75% to 94%, as assessed by chart review (for the period from recruitment to study completion at 6 months). To determine whether participation in the interventions leads to improvements in cancer treatment completion.

SECONDARY OUTCOMES:
Quality of life | 2 years
  The primary analytic approach for these secondary outcome variables will be a series of Linear Mixed-Effects Models (LMMS) modeling the change scores from baseline to each of the follow-up assessments, separately for each of the questionnaire outcome variables [51]. Analyses based on change scores have the advantage of creating easily interpretable results and clearly indicating the direction of individual change (e.g., increased protein intake).

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Gany, MD, MS, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (10):
- United States (10):
  - Brooklyn Hospital Center, Brooklyn, New York
  - Queens Hospital Center, Jamaica, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Bellevue Hospital Center, New York, New York
  - Ralph Lauren Center for Cancer Care and Prevention, New York, New York
  - St. Barnabas Medical Center, The Bronx, New York
  - Jacobi Medical Center, The Bronx, New York
  - Montefiore Health System (Montefiore Medical Center), The Bronx, New York
  - New York Cancer & Blood Specialists (Data collection only), The Bronx, New York
  - Lincoln Medical and Mental Health Center, The Bronx, New York

REFERENCES:
- [Derived] Gany F, Melnic I, Wu M, Li Y, Finik J, Ramirez J, Blinder V, Kemeny M, Guevara E, Hwang C, Leng J. Food to Overcome Outcomes Disparities: A Randomized Controlled Trial of Food Insecurity Interventions to Improve Cancer Outcomes. J Clin Oncol. 2022 Nov 1;40(31):3603-3612. doi: 10.1200/JCO.21.02400. Epub 2022 Jun 16. PMID 35709430
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/